CLINICAL TRIAL: NCT03765190
Title: A Phase I/II Study of Combination of Proton Therapy With Immunotherapy in Multiple Metastases Cancer
Brief Title: Combination of Proton Therapy With Immunotherapy in Multiple Metastases Cancer
Acronym: PI-MMC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: YiZhou International Cancer Hospital (Unknown)
Responsible Party: Principal Investigator, Xian-shu Gao, Professor, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20181204
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Proton Therapy; Immunotherapy; Neoplasm Metastasis
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Proton Therapy+PD-1 Ab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation: Proton Therapy+PD-1 Ab (Experimental): proton radiotherapy concurrent with immunotherapy(ie. PD-1 Ab for 1 year)
  Interventions: Combination Product: Radiation: Proton Therapy+PD-1 Ab

INTERVENTIONS:
Combination Product: Radiation: Proton Therapy+PD-1 Ab — combination of proton radiotherapy with PD-1 antibody

SUMMARY:
The purpose of this research study is to compare the effects (good and bad) on subjects and their cancer using proton radiation therapy in combination with immunotherapy(ie. Programmed cell death protein 1, also known as PD-1 antibody) in multiple metastases.

DETAILED DESCRIPTION:
As is known to all, the main treatment method for metastatic tumors is systemic chemotherapy and radiotherapy is merely for the purpose of palliative treatment. Recent studies have shown that tumors with no more than 5 metastatic sites can still achieve satisfactory overall survival by local treatments such as radiotherapy. However, for tumors with more metastatic lesions, side effect is pretty high for photon radiotherapy due to the wide range of irradiation. Protons might be a safe treatment means for multiple metastases cancer because of the Brag peak, when the normal tissue dose can be significantly reduced. Combination of proton therapy with immunotherapy can be a research direction for multiple metastatic tumors. This study intends to observe the safety and efficacy of proton technique combined with immunotherapy in improving the overall anti- tumor effect for metastatic tumors.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Unspecified Adult Solid Tumor
* Multiple metastatic tumors
* Intending to be treated with proton beam and immunotherapy
* Age ≥ 18 years old
* KPS≥70
* Signed written informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient under guardianship or tutorship
* Patients or legal guardians who are unable to understand informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Through 1 years after completion of treatment
  Assess adverse events according to CTCAE4.0

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Through 2 years after completion of treatment
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Overall survival (OS) | Through 2 years after completion of treatment
  OS is defined as the duration of time from start of treatment to time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Xianshu Gao, MD,PhD, Principal Investigator — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No